CLINICAL TRIAL: NCT06159439
Title: Validation of Contrast Enhanced Ultrasound (CEUS) for the Assessment of Renal Perfusion Using Renal Magnetic Resonance Imaging (MRI) in Chronic Kidney Disease (CKD
Brief Title: Establishing a New Ultrasound Technique to Improve Assessment of Chronic Kidney Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23018
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Chronic Kidney Diseases
Keywords: imaging; perfusion; contrast enhanced ultrasound
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with CKD having MRI and CEUS (Experimental): 10 participants with CKD will have an MRI scan and a contrast enhanced ultrasound scan. The two scans will be done within 7 days of each other.
  Interventions: Diagnostic Test: Contrast enhanced ultrasound scan; Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: Contrast enhanced ultrasound scan — Contrast enhanced ultrasound using Sonovue microbubble contrast
Diagnostic Test: MRI scan — Arterial-spin labelling magnetic resonance imaging

SUMMARY:
Blood flow to the kidneys is important in the development of kidney diseases. Currently we do not have ways of measuring and monitoring kidney blood flow for patients in real-time. This is a major barrier to investigation and management of acute kidney injury (AKI) and chronic kidney disease (CKD).

Kidney blood flow can be reliably measured using a specialised type of MRI scan, but this is expensive and difficult to do in people who are unwell. Contrast-enhanced ultrasound (CEUS) is a new technique, which uses a contrast containing microbubbles to measure blood flow. The benefits of this method are that it is relatively inexpensive, the contrast agents are not kidney-damaging and it can be done at the bedside.

We want to compare contrast enhanced ultrasound against the current best-measure of kidney blood flow, to see if it is giving accurate information about kidney blood flow. We will do this by doing both MRI and contrast enhanced ultrasound scans in people with chronic kidney disease and comparing the results.

DETAILED DESCRIPTION:
Renal perfusion, the delivery of oxygenated blood to kidney tissues, is relevant to a number of acute and chronic kidney diseases. Despite this, we do not have methods in current clinical practice to measure renal perfusion and monitor the response to supportive treatments in real time. This is a major barrier to investigation and management of acute kidney injury (AKI) and chronic kidney disease (CKD).

The current non-invasive gold standard technique for renal perfusion measurement is arterial-spin labelling magnetic resonance imaging (ASL-MRI), which has been validated against other measures of perfusion, including contrast agent-based methods. However, MRI has limitations including high cost, and logistical barriers. Therefore, validation of a bed-side measurement tool for renal perfusion would be of significant clinical importance.

This proposal aims to validate CEUS renal cortical perfusion measurement by comparison with quantifiable ASL-MRI parameters of renal microvascular perfusion in individuals with CKD.

TRIAL REGIMEN

All interventions outlined below are for the purposes of research, not usual care.

Study day:

All participants will attend fasted for preceding 2 hours. Demographic details and medical history will be recorded. The patient's concomitant medications which form part of their usual care will be recorded. These will not be adjusted.

Results of blood and urine tests that are collected as part of clinical care will be recorded.

Participants will undergo two scanning sessions, the first using renal MRI at the Sir Peter Mansfield Imaging Centre (SPMIC) to provide a quantitative measure of renal perfusion, and the second to provide the comparator measure of renal perfusion using CEUS performed at Royal Derby Hospital.

Outcomes:

MRI derived perfusion variables: peak time, and peak signal intensity (SI) will be obtained from time intensity curves.

Mean flow velocity (cm/s), cross-sectional area of the lumen (mm2), and hence bulk renal blood flow (ml/s)

CEUS derived perfusion parameters: acoustic index (AU); mean transit time (seconds); perfusion index, which is the ratio of AI to mTT; and wash-in rate (seconds)

ELIGIBILITY:
Inclusion Criteria:

* CKD 3b or CKD4
* Ability to give informed consent

Exclusion Criteria:

* Autosomal dominant polycystic kidney disease
* Solid organ transplant
* Pregnant women
* Known allergy to Sonovue
* Contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2025-02-02 (Estimated); Study Completion 2025-02-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between ASL-MRI measures of cortical perfusion (ml/ 100g/min) and CEUS measures of renal microvascular blood flow. | MRI scan and contrast enhanced ultrasound scan to be performed within 7 days of each other.
  The primary outcome will be the correlation between ASL-MRI measures of cortical perfusion (ml/ 100g/min) and CEUS measures of renal microvascular blood flow. As CEUS and ASL-MRI generate different units of measurement, correlations (rather than Bland-Altman analyses) will be used. We will define an ideal result as correlation coefficient r≥0.65, and adequate correlation coefficient r≥0.4.

SECONDARY OUTCOMES:
Repeatability of the CEUS measurements | 1 scan
  Repeatability of markers of perfusion between 5 flash-reperfusion sequences taken during 1 scan session
Correlation between global perfusion from PC-MRI corrected flow measures and CEUS | MRI scan and CEUS done within 7 days of each other
  As CEUS and ASL-MRI generate different units of measurement, correlations (rather than Bland-Altman analyses) will be used. We will define an ideal result as correlation coefficient r≥0.65, and adequate correlation coefficient r≥0.4.
Correlation between kinetic time-intensity parameters of CEUS and time-resolved MRA | MRI scan and CEUS done within 7 days of each other
  As CEUS and ASL-MRI generate different units of measurement, correlations (rather than Bland-Altman analyses) will be used. We will define an ideal result as correlation coefficient r≥0.65, and adequate correlation coefficient r≥0.4.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Selby, Principal Investigator — University of Nottingham

IPD SHARING:
Plan to Share IPD: No